CLINICAL TRIAL: NCT00932685
Title: Is Preoperative Distraction With a Hand Held Video Game Boy as Effective as Midazolam in Reducing Preoperative Anxiety Levels in Children as Weel as Emergence Agitation?
Brief Title: Does Distraction With a Hand Held Video Game Reduce Preoperative and Emergence Anxiety in Children?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Nintendo of North America (Unknown)
Responsible Party: Anuradha Patel, MD, University of Medicine & Dentistry of New Jersy
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0120030315A
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Pediatric Emergence Agitation and Pain
Keywords: pediatric emergence agitation and pain
MeSH Terms: conditions — Pain | interventions — Midazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2. Video Game (Active Comparator)
  Interventions: Device: Game Boy
- 1. Midazolam 0.5mg/kg (Active Comparator)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — Midazolam 0.5mg/kg
  Arms: 1. Midazolam 0.5mg/kg
Device: Game Boy — Children given video game as a distraction in preop holding and were permitted to continue playing the game in OR during induction
  Other Names: Nintendo-DS Game Boy
  Arms: 2. Video Game

SUMMARY:
Preoperative anxiety is characterized by subjective feelings of tension, apprehension, nervousness and worry. In children, preoperative anxiety is reported to result in postoperative negative psychological effects, including nightmares, eating problems and increased fear of doctors. Previous studies have assessed anxiety in children during the preoperative period and the effects of premedication and parental presence. Midazolzam has been shown to reduce preoperative anxiety in children but post operative recovery maybe delayed for children undergoing a short operative procedure. Distraction may be particularly helpful in children ages 6-12 as these children are curious about their environment. An association between preoperative anxiety and emergence agitation has been suggested. Emergence agitation in children is not well understood but is a frightening experience for child and parent. A previous study demonstrated the efficacy of hand held video games used as an interactive distraction to allay preoperative anxiety. The purpose of this study is to treat preop anxiety with premedication, or video game and to evaluate the impact of these interventions on the incidence and severity of emergence agitation.

ELIGIBILITY:
Inclusion Criteria:

* ASA rating of I-II Mask induction of General Anesthesia

Exclusion Criteria:

* Emergency surgery Children who have developmental disabilities or chronic illness Children who have had repetitive surgeries Children who have excessive anxiety attacks or who are currently on benzopaines

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2005-12; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
postoperative pain | on arrival in PACU, at 10 min, at 30 min and 10 minutes prior to discharge

SECONDARY OUTCOMES:
emergence agitation | on arrival, at 5 minutes and every 10 min for one hour in PACU

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Patel, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- University Hospital, Newark, New Jersey, United States